CLINICAL TRIAL: NCT00871468
Title: Does Anterior-Inferior Clavicle Plating Have a Lower Rate of Soft Tissue Irritation Compared to Superior Plating? A Prospective Randomized Trial
Brief Title: Plating Clavicle Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: United States Army Institute of Surgical Research (U.S. Federal Agency)
Collaborators: William Beaumont Army Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-08-003
Record Dates: First submitted 2009-03-26; First posted 2009-03-30 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2016-12

CONDITIONS: Clavicle Fracture, Non Union/Malunion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- superior plate (Active Comparator): Clavicle plate on the superior surface of the bone
  Interventions: Procedure: superior plate
- anterior inferior plate (Experimental): plate placed on anterior inferior surface of bone
  Interventions: Procedure: anterior-inferior plate

INTERVENTIONS:
Procedure: superior plate — Open reduction internal fixation (ORIF) clavicle with superior plate
  Arms: superior plate
Procedure: anterior-inferior plate — ORIF clavicle with anterior inferior plate
  Arms: anterior inferior plate

SUMMARY:
The anterior-inferior clavicle plate position will have a lower rate of soft tissue irritation that limits activity and/or requires hardware removal compared to superior plate position.

DETAILED DESCRIPTION:
Compare the rates of soft-tissue irritation with two different methods of plating for clavicle fractures. Patients will be randomized to anterior-inferior or superior plating. Validated shoulder scoring systems will be used to assess outcome. Specific follow-up questions will address the patient's ability to wear his/her uniform, body armor, ruck sack, and other shoulder-borne equipment over the surgical site.

ELIGIBILITY:
Inclusion Criteria:

* Active duty, Reservists, National Guard service members
* completely displaced shaft fracture of the clavicle (no cortical contact between the main proximal and distal fragments)
* a fracture involving the middle third of the clavicle (a fracture amenable to plate fixation with a minimum of three screws in each proximal and distal fragment)
* chronic nonunion and malunion fractures
* no medical contraindications to general anesthesia
* provided informed consent.

Exclusion Criteria:

* an age of less than eighteen years or greater than sixty five years
* a fracture in the proximal or distal third of the clavicle not amenable to plating
* a pathological fracture
* an associated head injury (a Glasgow Coma Scale score of <15 at 21 days after injury)
* an inability to comply with followup
* a medical contraindication to surgery and/or anesthesia (such as heart disease, renal failure, or active chemotherapy)
* a lack of consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2008-10; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Less irritation with anterior-inferior plating and less need for hardware removal. | 2 years

SECONDARY OUTCOMES:
DASH (Disability of Arm, Shoulder and Hand) and constant scores | 2 years

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - William Beaumont Army Medical Center, El Paso, Texas
  - US Army Institute of Surgical Research, Fort Sam Houston, Texas